CLINICAL TRIAL: NCT00001840
Title: Evaluation of Treated and Untreated Stroke
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990041; 99-CC-0041
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-01

CONDITIONS: Cerebrovascular Accident; Infarction; Ischemia
Keywords: Infarct; Ischemia; MRI; Natural History; Stroke; Treatment; Brain Stroke
MeSH Terms: conditions — Stroke; Infarction; Ischemia

SUMMARY:
This project will investigate the evolution of treated and untreated stroke in patients recruited from the collaborative brain stroke program between NINDS, CC, and Suburban Hospital. The study will use anatomical and functional imaging techniques with emphasis on the acute and subacute stage (less than one month) of the disease.

As the availability of new therapeutic options for the management of acute brain stroke increases, the need to define the evolution of the disease becomes paramount, particularly as therapeutic windows, defined by known and perhaps yet undiscovered parameters, may exist. Defining these parameters will be based on state-of-the-art imaging technology with the potential of clarifying the division between ischemia (reversible damage) and infarction (irreversible). Measures of lesion size and distribution along with vascular morphology, diffusion, perfusion, flow-related, and metabolic measures will be obtained over time. We foresee these measurements will significantly develop our understanding of cerebral ischemia and introduce diagnostic and quantitative tools to guide therapy and measure its efficacy.

DETAILED DESCRIPTION:
This project will investigate the evolution of treated and untreated stroke in patients recruited from the collaborative brain stroke program between NINDS, CC, and Suburban Hospital. The study will use anatomical and functional imaging techniques with emphasis on the acute and subacute stage (less than one month) of the disease.

As the availability of new therapeutic options for the management of acute brain stroke increases, the need to define the evolution of the disease becomes paramount, particularly as therapeutic windows, defined by known and perhaps yet undiscovered parameters, may exist. Defining these parameters will be based on state-of-the-art imaging technology with the potential of clarifying the division between ischemia (reversible damage) and infarction (irreversible). Measures of lesion size and distribution along with vascular morphology, diffusion, perfusion, flow-related, and metabolic measures will be obtained over time. We foresee these measurements will significantly improve our understanding of cerebral ischemia and introduce diagnostic and quantitative tools to guide therapy and measure its efficacy.

ELIGIBILITY:
Any subject suspected of having a stroke based on the NIH Stroke Scale and age 21 years or over.

Subjects will be enrolled into this protocol only if they are determined intellectually capable of providing their own informed consent.

No subjects will be included if they have a condition which would preclude their entry into the scanner (e.g., paralyzed hemidiaphragm, morbid obesity, claustrophobia, etc.) or present unnecessary risks (e.g., surgery of uncertain type, symptoms of pheochromocytoma or insulinoma, etc.).

No women who are pregnant or lactating.

No subjects with hemoglobinopathies and asthma.

No subjects with renal or hepatic disease.

No subjects who have a contraindication to MR scanning such as surgery that involves metal clips or wires which might be expected to concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field (e.g., aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or autodefibrillator, cochlear implant, ocular foreign body and mechanical pump).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1999-02; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wolpert SM, Bruckmann H, Greenlee R, Wechsler L, Pessin MS, del Zoppo GJ. Neuroradiologic evaluation of patients with acute stroke treated with recombinant tissue plasminogen activator. The rt-PA Acute Stroke Study Group. AJNR Am J Neuroradiol. 1993 Jan-Feb;14(1):3-13. PMID 8427107
- [Background] Hossmann KA. Viability thresholds and the penumbra of focal ischemia. Ann Neurol. 1994 Oct;36(4):557-65. doi: 10.1002/ana.410360404. PMID 7944288
- [Background] Bryan RN, Levy LM, Whitlow WD, Killian JM, Preziosi TJ, Rosario JA. Diagnosis of acute cerebral infarction: comparison of CT and MR imaging. AJNR Am J Neuroradiol. 1991 Jul-Aug;12(4):611-20. PMID 1688347